CLINICAL TRIAL: NCT04285866
Title: Spanish Real World Data on Unresectable Stage III NSCLC Patients Treated With Durvalumab After Chemoradiotherapy.
Brief Title: Spanish Real World Data on Patients Treated With Durvalumab After Chemoradiotherapy.
Acronym: S-REAL
Status: Completed | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 19/02_S-REAL
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Locally advanced small cell lung cancer; SCLC; lung cancer; durvalumab after chemotherapy; real world data
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Durvalumab Group: Patients who have participated in the EAP between 1 September 2017 up to 21 December 2018 and have received at least 1 dose of durvalumab.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab after chemoradiotherapy
  Other Names: MEDI4736

SUMMARY:
This is a non-interventional, observational, multicentre, one-arm, non-comparative, and retrospective study.

The study is based on the collection of data about the patients treated with Durvalumab after chemoraditherapy in the real world. The patients participating in this non-interventional study will not receive treatment in relation to the study. The primary objective is to assess affectiveness of durvalumab in patients treated in real-life settings by evaluating Progression Free Survival.

DETAILED DESCRIPTION:
Lung Cancer represent approximately 13% of total cancer diagnoses worldwide and continues to be the leading cause of cancer-related mortality. Stage III represents between 25-30% of NSCLC and the majority of them are unresectable. The standard treatment in unresectable patients was chemoradiotherapy consurrently if possible.

The PACIFIC study is a phase III study to evaluate the efficacy and safety of durvalumab as a sequential therapy concurrent platinum-based chemotherapy and thoracic RT. The study was positive for both primary endpoints progression-free survival and overall survival. After that, it was decided to open an early acces programme ti provide acces to durvalumab for patients with locally advanced, unresectable NSCLC (stage III) tho have not progressed following chemoradiation.

This observational study is based on the collection of data about the patients treated with Durvalumab after chemoraditherapy in the real world.

The study will include all patients who have participated in the EAP between 1 September 2017 up to 21 December 2018 and have received at least 1 dose of durvalumab.

The primary objective is to assess affectiveness of durvalumab in patients treated in real-life settings by evaluating Progression Free Survival. Other secondary objectives are:

To assess effectiveness of durvalumab in patients treated in real-life settings by evaluating 1-year survival rate, to describe adverse events of special interests, to stimate time and sites of disease progression or relapse in metastatic setting, to describe details on durvalumab treatment, to describe demographic and clinical characteristics of stage III unresectable NSCLC patients treated with Durvalumab, to describe previous chemoradiotherapy strategy, to describe the baseline staging status, to further assess subsequent treatments pattern at the time of disease progression including duration of therapy and type of therapy, and to explore healthcare resource utilization while on durvalumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically documented diagnosis of NSCLC with a locally advanced, or locally recurrent, unresectable (stage III) disease (according to American Joint Committee on Cancer [AJCC] lung cancer edition 7 or 8).
2. Age ≥ 18 years at time of study Entry
3. Patients must have been treated with chemotherapy and radiotherapy concurrently or sequentially and shown no progressive disease following chemoradiation
4. Patients must have been enrolled in durvalumab EAPs between 1 September 2017 and 21 December 2018.
5. Patients must have been treated with at least one dose of durvalumab within the EAP
6. Alive patients must have signed, dated and IRB/EC-approved written informed consent* form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.

Exclusion Criteria:

1. Alive patients who do not want to sign and date an IRB/IEC-approved written informed consent form.
2. Patients who were accepted in the EAP, but did not receive treatment.
3. Patients treated with durvalumab in clinical studies prior to the index date (first dose of durvalumab received within the EAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have parcipated in the EAP between 1 September 2017 up to 21 December 2018 and have received at least 1 dose of durvalumab.
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of the first dose of durvalumab received (within the EAP) to the date of disease progression, death, or the end of follow-up, assessed up to 60 months
  To assess effectiveness of durvalumab in patients treated in real-life settings by evaluating PFS

SECONDARY OUTCOMES:
1-year survival rate | 1 year
  To assess effectiveness of durvalumab in patients treated in real-life settings by evaluating 1-year survival rate.
To describe adverse events of special interest (AESIs) | From date of the first dose of durvalumab received (within the EAP) to the date of disease progression, death, or the end of follow-up, assessed up to 60 months
  To describe AESIs leading to treatment temporary interruption or permanent discontinuation of durvalumab, or which require interventions of concomitant use of corticosteroids, immunosupressants and/or endocrine therapies.
Time and site of disease progression or relapse | From date of the first dose of durvalumab received to the date of disease progression, assessed up to 60 months
  To estimate time and sites of disease progression or relapse in metastatic setting.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Garrido, MD, Study Chair — Fundación GECP Investigator
Locations (39):
- Spain (39):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Costa del Sol, Marbella, Málaga
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitario De La Ribera, Alzira, Valencia
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital de A Coruña, A Coruña
  - Hospital General de Alicante, Alicante
  - Consorci Mar Parc de Salut de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital de Sanchinarro, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Complexo Hospitalario de Ourense, Ourense
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital General de Segovia, Segovia
  - Hospital Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitari i Politécnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org